CLINICAL TRIAL: NCT02829021
Title: Dynamic Infrared Thermography in Breast Cancer Diagnostics. A Diagnostic Accuracy Study Comparing Dynamic Infrared Thermography Against Mammography (Reference Standard)
Brief Title: Dynamic Infrared Thermography in Breast Cancer Diagnostics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of North Norway (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: REK-109/2008; FAST-67 (Registry Identifier: University hospital of North Norway)
Record Dates: First submitted 2016-04-12; First posted 2016-07-12 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2016-06

CONDITIONS: Breast Cancer
Keywords: Sensitivity; Specificity; Breast cancer; Mammography; Thermography; Infrared; Dynamic; Diagnostic accuracy; Diagnostic odds ratio
MeSH Terms: conditions — Breast Neoplasms; Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Thermography and mammography (Other): All participants will be examined with
  1. Dynamic infrared thermography (FLIR ThermaCAM P-65)
  2. Mammography, clinical examination and if necessary breast tissue biopsy to diagnose breast cancer.
  Interventions: Device: FLIR ThermaCAM P-65

INTERVENTIONS:
Device: FLIR ThermaCAM P-65 — Women recalled for assessment after positive screening mammography were offered dynamic infrared thermography before clinical mammography and further tests.
  Other Names: Serial number: 25300659

SUMMARY:
This study evaluate diagnostic accuracy of dynamic infrared thermography compared to mammography (reference test) in breast cancer diagnostics. Women aged 50-70 years, selected for assessment after mammography screening were invited to dynamic infrared thermography before clinical mammography and further examination.

DETAILED DESCRIPTION:
This study evaluate diagnostic accuracy of dynamic infrared thermography compared to mammography (reference test) in breast cancer diagnostics.

Dynamic infrared thermography (DIRT) is an imagine procedure offering a non-invasive, painless examination without risk of radiation. Dynamic infrared thermography does not provide information on the morphological characteristics of the breast, rather it provides functional information on thermal and vascular conditions of the tissue (Fitzgerald, 2012).

During the study period from April 2009 until June 2012, a total of 168 women aged 50-70 years who were recalled for assessment after positive mammography screening were offered dynamic infrared thermography before further tests (clinical mammography, clinical examination and if necessary breast tissue biopsy).

Radiographers at the Breast Diagnostic Center (BDS) at University Hospital North Norway collected information about parity, menopausal status, use of hormone therapy and size of bra.

The same radiographers also carried out all the dynamic infrared thermography examinations. PI Åshild O. Miland and Professor James B. Mercer interpreted the thermograms and entered the data into the thermography database. Both were blinded for further assessments (mammography, clinical examination and biopsy) and non of them talked to any of the participants after the examination.

The health professionals who were responsible for the women during mammography, clinical examination and biopsy were blinded for the results from the infrared digital thermography examination. They were not allowed to ask the women about the infrared digital thermography examination.

The three radiologists at BDS made the interpretation of the mammographies and entered data into the digital patient journal and to the mammography database at The Norwegian Cancer Registry. One of the radiologist took, when necessary, breast biopsies. A breast surgeons were responsible for the clinical breast examination. Pathologists verified the histology.

Breast radiologist Jan Ole Frantzen and researcher Merethe Kumle, MD, PhD collected information about breast cancer results from the digital patient journal and Roentgen information system (RIS) and entered it into a separate mammography database.

The thermography database and the mammography database was still not merged at the time of registration in ClinicalTrials.gov (March 2015).

ELIGIBILITY:
Inclusion Criteria:

* women,
* aged 50-69
* attending the Norwegian Breast Screening Program,
* recalled for assessment after positive mammography screening

Exclusion Criteria:

* not attending the Norwegian Breast Screening Program,
* recalled to mammography for other reason than positive screening mammogram.

Ages: 50 Years to 69 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2009-04; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy of Thermography compared with Mammography and breast biopsy. | Baseline
  Can thermography distinguish benign from malign tumours in breast cancer diagnostics. The gold standard is breast biopsy pathology.
  The outcome is measured as number of subjects with pathological diagnosis of cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Åshild O. Miland, PhD, Principal Investigator — Senior lecturer
Locations (1):
- Åshild Odden Miland, Tromsø, Tromsø, Norway

IPD SHARING:
Plan to Share IPD: Undecided
This is a small Diagnostic Accuracy Study, the investigators will decide upon data sharing when they have finished the statistical analysis. If someone is interested in the data, please contact the investigators.